CLINICAL TRIAL: NCT00598741
Title: Dynamic Contrast Enhanced MRI(DCE-MRI)of Bone Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other); University of Oregon (Other); University College, London (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-083
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Sarcoma; Bone Tumor
Keywords: Bone; Sarcoma; 04-083
MeSH Terms: conditions — Sarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: DCE-MRI

INTERVENTIONS:
Other: DCE-MRI — Patients will undergo DCE-MRI prior to, and within 18-24 days of starting chemotherapy. These studies are designed to determine if the DCE-MRI data will provide an a priori or early prognostic marker of tumor response. The dynamic MRI is done on a standard clinical scanner using standard techniques described below.
  MR imaging studies will be acquired on a 1.5T GE (Milwaukee,WI) Signa LX scanner.

SUMMARY:
The purpose of this study is to see whether fast imaging with MRI and the usual contrast material used for MRI, predicts which patients will do well with treatment. Some studies suggest that MRIs done right before surgery may be able to tell how much of the cancer was killed by the chemotherapy. This study will see if this is true in patients with osteogenic sarcoma (OS) and Ewing's sarcoma (ES). This study will also see if MRIs done early in treatment can tell if the chemotherapy is working.

DETAILED DESCRIPTION:
Patients will undergo DCE-MRI studies prior to chemotherapy, 18-24 days after starting treatment, continue treatment and undergo a third MRI within 25 days prior to surgery. All patients with OS or Ewing sarcoma who will undergo pre-operative chemotherapy are eligible for study. Anti-neoplastic therapy will be determined by the primary physician and will not be impacted upon by this study, although the data will be made available to the physicians involved in the patient's care. The goals of this study are: 1) To determine if pre-operative dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) can reliably predict percent necrosis at definitive surgery in bone tumors after induction chemotherapy. 2) Evaluate the hypothesis that in patients with Ewing or osteogenic sarcoma (OS), the a priori or early (18-24 days into treatment) DCE-MRI study predicts pathological percent necrosis measured at surgery, and disease free survival. 3) Determine if the DCE-MRI results are independent markers of tumor response compared to current clinical markers (LDH, alkaline phosphatase (osteogenic sarcoma only), primary disease site, primary disease size (length and volume), stage). 4) Compare the DCE-MRI results with several key molecular parameters including p53 mutations and CDKN2A deletion in Ewing's sarcoma and RB alterations, CDKN2A deletion, and expression of HER-2, platelet derived growth factor, reduced folate carrier, and pglycoprotein in osteogenic sarcoma. Ewing's sarcoma and osteogenic sarcoma samples will also be submitted for Affymetrix expression microarray analysis. Summary: This project will determine the potential of DCE-MRI to predict tumor necrosis and as an a priori or early marker of tumor response to neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologically proven diagnoses of OS or Ewing Sarcoma undergoing induction chemotherapy are eligible for study.
* Patients/guardians must provide written consent. It is anticipated that many of these patients will be minors and consent will be obtained from their parent/guardian.
* The presence of the evaluable primary tumor is required.

Exclusion Criteria:

* Inability to cooperate for an MRI.
* Absence of evaluable primary tumor
* Known reaction to Gd-DTPA
* Pre-operative radiation to primary tumor site
* Contraindication to MRI

  1. Pacemaker
  2. Aneurysmal clips
  3. Metal implants in field of view
  4. Any other conditions that result in patients not being appropriate for MRI. study
  5. Pregnancy
  6. Age and mental status wherein he/she is able to cooperate for MRI study
  7. Unusual histopathologic subvariants (radiation induced, Paget's disease, hereditary RB)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pts will undergo baseline MRI prior to begin chemotherapy. Bet 18-24 days after beginning chemotherapy, they will undergo second MRI. They will continue chemotherapy and w/in 25 days prior definitive surgery, will undergo another MRI. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Koutcher, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org